CLINICAL TRIAL: NCT00679354
Title: Cilengitide (EMD 121974) (IND# 59073) in Recurrent or Progressive and Refractory Childhood High-Grade Glioma
Brief Title: Cilengitide in Treating Younger Patients With Recurrent or Progressive High-Grade Glioma That Has Not Responded to Standard Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00339; NCI-2009-00339 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ACNS0621; CDR0000595623; ACNS0621 (Other: Children's Oncology Group); ACNS0621 (Other: CTEP); U10CA098543 (NIH); NCT01648400 (obsolete NCT alias)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Recurrent Childhood Anaplastic Astrocytoma; Recurrent Childhood Anaplastic Oligoastrocytoma; Recurrent Childhood Anaplastic Oligodendroglioma; Recurrent Childhood Brain Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Glioblastoma; Recurrent Childhood Visual Pathway and Hypothalamic Glioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Optic Nerve Glioma | interventions — Cilengitide

ARMS (1):
- Treatment (cilengitide) (Experimental): Patients receive cilengitide IV over 1 hour on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cilengitide; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial studies how well cilengitide works in treating younger patients with recurrent or progressive high-grade glioma that has not responded to standard therapy. Cilengitide may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate to cilengitide in younger patients with recurrent or progressive high-grade glioma that is refractory to standard therapy.

SECONDARY OBJECTIVES:

I. To estimate the distribution of time to progression, time to treatment failure, and time to death in these patients.

II. To estimate the rate of toxicity, especially symptomatic intratumoral hemorrhage, in these patients.

III. To evaluate the pharmacokinetics of cilengitide in plasma using a limited sampling strategy.

IV. To evaluate the pharmacogenetic polymorphisms in drug transporters (eg, breast cancer resistance protein [BCRP], P-glycoprotein [P-gp]) and relate to cilengitide disposition.

OUTLINE:

Patients receive cilengitide IV over 1 hour on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary central nervous system (CNS) high-grade glioma, including any of the following:

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * High-grade astrocytoma not otherwise specified (i.e., anaplastic ganglioglioma, anaplastic mixed glioma, or anaplastic mixed glioneuronal tumors)

    * No diffuse pontine gliomas, gliomatosis cerebri, and primary spinal cord high-grade astrocytoma
  * Gliosarcoma
* Recurrent or progressive disease that is refractory to standard therapy
* Radiographically documented measurable disease

  * Lesion must be at least twice the thickness of the image from which it is derived (e.g., 10 mm for a 5 mm slice thickness)
* No diffuse pontine gliomas
* No evidence of prior CNS bleeding
* Karnofsky performance status (PS) 50-100% (patients > 16 years of age)
* Lansky PS 50-100% (patients =< 16 years of age)
* Life expectancy >= 8 weeks
* Absolute neutrophil count (ANC) >= 1,000/μL
* Platelet count >= 100,000/μL (transfusion independent)
* Hemoglobin >= 8.0 g/dL (red blood cell [RBC] transfusions allowed)
* Creatinine clearance or radioisotope glomerular filtration rate >= 70mL/min OR serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4mg/dL (female) (>= 16 years of age)
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 times ULN for age
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94%, if determination is clinically indicated
* Seizure disorder is allowed provided it is well-controlled with anticonvulsants
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Recovered from all prior therapy
* No more than two prior treatments for high-grade glioma (i.e., one initial treatment and one treatment for relapse)
* More than 2 weeks since prior myelosuppressive chemotherapy (>= 6 weeks for nitrosoureas)
* At least 1 week since prior non-myelosuppressive chemotherapy, immunotherapy, or biologic therapy
* At least 2 weeks since prior local palliative radiotherapy (i.e., small port) to a symptomatic non-target lesion only
* At least 3 months since prior craniospinal radiotherapy
* At least 6 weeks since prior substantial bone marrow radiotherapy
* At least 6 months since prior allogeneic stem cell transplant (SCT) or rescue

  * Patients who have undergone prior allogeneic SCT and who have graft-versus-host disease (GVHD) must have controlled GVHD that is =< grade 2
* At least 1 month since prior autologous SCT
* More than 1 week since prior growth factors (> 3 weeks for pegfilgrastim [Neulasta®])
* No other concurrent anticancer therapy, including chemotherapy or immunomodulating agents
* No other concurrent experimental agents or therapies
* No concurrent alternative or complimentary therapies
* No concurrent homeopathic medicines
* No concurrent nonsteroidal anti-inflammatory drugs (NSAIDs) or acetylsalicylic acid (aspirin)
* No concurrent steroids as anti-emetics
* Concurrent steroids for treatment of increased intracranial pressure allowed if on a stable or decreasing dose for >= 1 week before study entry
* Concurrent radiotherapy to localized painful lesions allowed provided >= 1 measurable lesion is not irradiated

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobey MacDonald, Principal Investigator — Children's Oncology Group
Locations (20):
- United States (19):
  - Kaiser Permanente-Oakland, Oakland, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York University Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cilengitide): Patients receive cilengitide IV over 1 hour (1800 mg/m2/dose, maximum 75mg/kg) on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Cilengitide)
Started | 30
Completed | 0
Not Completed | 30
Not completed — Death | 3
Not completed — Lack of Efficacy | 22
Not completed — Physician Decision | 4
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 13 [1 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 20
  More than one race | 0
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 28
  Canada | 1
  Australia | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response to Cilengitide
Description: Objective response is defined as a complete response or partial response at 4 weeks that is sustained for at least another 4 weeks, or a stable disease at 4 weeks that is sustained for at least 12 weeks while on stable or decreasing dose of corticosteroids, except when corticosteroids are being used to control hydrocephaly unrelated to tumor progression.
Time Frame: Up to 16 weeks
Population: Six patients are considered inevaluable for objective response (including one ineligible patient) and excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 24
participants
  With Objective Response | 1
  Without Objective Response | 23

2. Secondary Outcome: Time to Tumor Progression (TTP)
Description: The distribution of TTP will be analyzed separately using product limit (PL) estimate.
Time Frame: Time from study enrollment to radiographically determined tumor progression or recurrence, assessed up to 5 years
Population: 29 eligible patients are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 29
Days | 28 [25 to 41]

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: The distribution of TTF will be analyzed separately using PL estimate.
Time Frame: Time from study enrollment to tumor progression, tumor recurrence, death from any cause, or occurrence of a second malignant neoplasm, assessed up to 5 years
Population: Twenty-nine eligible patients are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 29
Days | 28 [25 to 41]

4. Secondary Outcome: Time to Death (TTD)
Description: The distribution of TTD will be analyzed separately using PL estimate.
Time Frame: Time from study enrollment to death from any cause, assessed up to 5 years
Population: Twenty-nine eligible patients are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 29
Days | 172 [99 to 226]

5. Secondary Outcome: Rate of Toxicity, Especially That of Symptomatic Intratumoral Hemorrhage (ITH) Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Description: Rate of individual toxicity including that of symptomatic ITH will be summarized in each course of treatment using standard descriptive statistical methods.
Time Frame: Up to 5 years
Population: Twenty-nine eligible patients are included in the analysis. One patient was excluded due to ineligibility.
Measure: Number; unit: percent of pts with symptomatic ITH
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 29
percent of pts with symptomatic ITH | 6.9

6. Secondary Outcome: Pharmacokinetic Parameter of Cilengitide in Plasma: Volume of Central Compartment (Vc)
Description: Cilengitide plasma concentration-time data are fit to a compartmental pharmacokinetic model using MAP-Bayesian estimation as implemented in ADAPT II. For each patient, samples collected at different time points are used to derive one Vc value per patient.
Time Frame: At baseline and 1, 3, and 6 hours after the first dose of cilengitide
Population: All 18 patients consenting for pharmacokinetic study are included in this analysis.
Measure: Median (Full Range); unit: L/m^2
Groups:
- Treatment (Cilengitide): Patients receive cilengitide IV over 1 hour (1800 mg/m2/dose, maximum 75mg/kg) on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 18
L/m^2 | 6.20 [3.34 to 10.72]

7. Secondary Outcome: Pharmacokinetic Parameter of Cilengitide in Plasma: Elimination Rate Constant (Ke)
Description: Cilengitide plasma concentration-time data are fit to a compartmental pharmacokinetic model using MAP-Bayesian estimation as implemented in ADAPT II. For each patient, samples collected at different time points are used to derive one Ke value per patient.
Time Frame: At baseline and 1, 3, and 6 hours after the first dose of cilengitide
Population: All 18 patients consenting for pharmacokinetic study are included in this analysis.
Measure: Median (Full Range); unit: hr^(-1)
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 18
hr^(-1) | 0.58 [0.36 to 1.00]

8. Secondary Outcome: Pharmacokinetic Parameter of Cilengitide in Plasma: Half-life (t1/2)
Description: Cilengitide plasma concentration-time data are fit to a compartmental pharmacokinetic model using MAP-Bayesian estimation as implemented in ADAPT II. For each patient, samples collected at different time points are used to derive one t1/2 value per patient.
Time Frame: At baseline and 1, 3, and 6 hours after the first dose of cilengitide
Population: All 18 patients consenting for pharmacokinetic study are included in this analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 18
hours | 1.26 [0.69 to 1.90]

9. Secondary Outcome: Pharmacokinetic Parameter of Cilengitide in Plasma: Systemic Clearance (Cl)
Description: Cilengitide plasma concentration-time data are fit to a compartmental pharmacokinetic model using MAP-Bayesian estimation as implemented in ADAPT II. For each patient, samples collected at different time points are used to derive one Cl value per patient.
Time Frame: At baseline and 1, 3, and 6 hours after the first dose of cilengitide
Population: All 18 patients consenting for pharmacokinetic study are included in this analysis.
Measure: Median (Full Range); unit: L/hr/m^2
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 18
L/hr/m^2 | 3.84 [2.47 to 5.75]

10. Secondary Outcome: Pharmacogenetic Polymorphism in Drug Transporter Gene ABCB1 and Relate to Cilengitide Disposition as Measured by AUC
Description: Cilengitide systemic exposure as measured by AUC is used in this genotype-phenotype analysis. The ABCB1 (P-glycoprotein; P-gp) Exon 26 genotype is coded as 0/1/2 based on the number of T alleles.
Time Frame: At baseline
Population: The analysis includes 12 eligible patients with both AUC data and ABCB1 Exon 26 data available.
Measure: Number; unit: Spearman's correlation
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 12
Spearman's correlation | 0.00
Statistical Analysis 1: Comparison: Treatment (Cilengitide); Test type: Superiority or Other; p = 1.000, Spearman's Correlation; Spearman's Correlation Coefficient = 0.00

11. Secondary Outcome: Pharmacogenetic Polymorphism in Drug Transporter Gene ABCB1 and Relate to Cilengitide Disposition as Measured by Systemic Clearance
Description: Cilengitide systemic exposure as measured by systemic clearance is used in this genotype-phenotype analysis. The ABCB1 (P-glycoprotein; P-gp) Exon 26 genotype is coded as 0/1/2 based on the number of T alleles.
Time Frame: At Baseline
Population: The analysis includes 12 eligible patients with both systemic clearance data and ABCB1 Exon 26 data available.
Measure: Number; unit: Spearman's Correlation
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 12
Spearman's Correlation | 0.56
Statistical Analysis 1: Comparison: Treatment (Cilengitide); Test type: Superiority or Other; p = 0.057, Spearman's Correlation; Spearman's Correlation Coefficient = 0.56

12. Secondary Outcome: Pharmacogenetic Polymorphism in Drug Transporter Gene ABCG2 and Relate to Cilengitide Disposition as Measured by AUC
Description: Cilengitide systemic exposure as measured by AUC is used in this genotype-phenotype analysis. The ABCG2 (breast cancer resistance protein; BCRP) Exon 5 genotype is coded as 0/1/2 based on the number of G alleles.
Time Frame: At baseline
Population: The analysis includes 12 eligible patients with both AUC data and ABCG2 Exon 5 data available.
Measure: Number; unit: Spearman's Correlation
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 12
Spearman's Correlation | -0.22
Statistical Analysis 1: Comparison: Treatment (Cilengitide); Test type: Superiority or Other; p = 0.495, Spearman's Correlation; Spearman's Correlation Coefficient = -0.22

13. Secondary Outcome: Pharmacogenetic Polymorphism in Drug Transporter Gene ABCG2 and Relate to Cilengitide Disposition as Measured by Systemic Clearance
Description: Cilengitide systemic exposure as measured by systemic clearance is used in this genotype-phenotype analysis. The ABCG2 (breast cancer resistance protein; BCRP) Exon 5 genotype is coded as 0/1/2 based on the number of G alleles.
Time Frame: At baseline
Population: The analysis includes 12 eligible patients with both systemic clearance data and ABCG2 Exon 5 data available.
Measure: Number; unit: Spearman's Correlation
Arm/Group | Treatment (Cilengitide)
Number analyzed (Participants) | 12
Spearman's Correlation | -0.48
Statistical Analysis 1: Comparison: Treatment (Cilengitide); Test type: Superiority or Other; p = 0.114, Spearman's Correlation; Spearman's Correlation Coefficient = -0.48

ADVERSE EVENTS:
Description: Only eligible patients are included in the Toxicity reporting for both Serious and Other AEs. One patient was excluded from AE reporting because patient was deemed ineligible.
Arm/Group | Treatment (Cilengitide)
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 8/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cilengitide) (N=29)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Death NOS (General disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Fever (General disorders) | 1
Headache (Nervous system disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cilengitide) (N=29)
Allergic reaction (Immune system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Headache (Nervous system disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary incontinence (Renal and urinary disorders) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less